CLINICAL TRIAL: NCT01724853
Title: Outcomes of Treatment for Trapeziometacarpal Osteoarthritis Using a Comprehensive Core Set.
Brief Title: Outcomes of Treatment for Trapeziometacarpal Osteoarthritis
Acronym: RASSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Herren, MD, MHA, Schulthess Klinik
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: RASSH01
Record Dates: First submitted 2012-11-01; First posted 2012-11-12 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthrosis of the Carpometacarpal Joint of the Thumb
Keywords: Carpometacarpal; osteoarthritis; outcome measures
MeSH Terms: conditions — Osteoarthritis | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Other): Preferred surgery
  Interventions: Procedure: Surgery
- Conservative (Other): Conservative treatment
  Interventions: Other: Conservative

INTERVENTIONS:
Procedure: Surgery — Resection suspension interposition arthroplasty or Arthrodesis
  Arms: Surgery
Other: Conservative — Injection
  Arms: Conservative

SUMMARY:
The main objective of the study is the evaluation of the outcomes following treatment for TMC OA using a set of variables covering all OMERACT categories as well as the dimensions of the International Classification of Functioning, Disability and Health (ICF). Secondary aims are the analysis of the determinants of patient satisfaction with the treatment result, the evaluation of the psychometric properties of the Michigan Hand Outcomes Questionnaire (MHQ), which has not yet been established in TMC OA patients, as well as the economic impact associated with TMC OA.

DETAILED DESCRIPTION:
Hand osteoarthritis is a frequent condition in the middle-aged and elderly population with a prevalence of up to 76%. After the distal interphalangeal joints, the trapeziometacarpal joints are the most affected joints of the hand. Symptoms such as pain, stiffness, deformity, loss of grip strength, as well as reduction of joint mobility, are affecting the overall hand function and patients' quality of life. Numerous studies have evaluated different surgical and conservative interventions for treating patients with trapeziometacarpal osteoarthritis (TMC OA) with both interventions found to be effective in reducing pain and increasing function. To date, there is only little evidence about the characteristics and outcomes of patients who receive a conservative or a surgical treatment for TMC OA. The analysis should focus on which factors contribute to either a conservative or a surgical treatment, and if these patients differ regarding personal or health-related factors. Furthermore, no data about the economic consequences of a resection interposition suspension arthroplasty are available which highlights the need for a financial analysis of this procedure with respect to the benefit for the patient and cost bearers.

Besides objective parameters, such as strength and range of motion, the evaluation of patient satisfaction as well as the fulfilment of preoperative expectation is becoming increasingly important as outcome measures. However, there is no standardized instrument available for measuring satisfaction, expectations and their fulfillment for TMC OA patients.

For measuring outcomes of OA, a core set for outcome measures for OA trials (hip, knee, hand) was developed at the OMERACT III conference. It comprised of the assessment of pain, physical function, patients' global condition and joint imaging. Furthermore, the evaluation of quality of life is recommended, but the specific items of this core set for TMC OA patients still remain to be defined.

The main objective of the study is the evaluation of the outcomes following treatment for TMC OA using a set of variables covering all OMERACT categories as well as the dimensions of the International Classification of Functioning, Disability and Health (ICF). Secondary aims are the analysis of the determinants of patient satisfaction with the treatment result, the evaluation of the psychometric properties of the Michigan Hand Outcomes Questionnaire (MHQ), which has not yet been established in TMC OA patients, as well as the economic impact associated with TMC OA.

In order to achieve these objectives, a prospective cohort study including patients with TMC OA will be conducted, regardless of if they will have surgery or not. A total of 100 surgically treated patients will be analysed during a one-year inclusion period and all conservatively treated patients will also be analysed during the same time. Follow up examinations will take place at 3, 6 and 12 months for all patients using a standardized set of objective as well as subjective outcome measurements including the MHQ.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients diagnosed for TMC OA
* signed informed consent

Exclusion Criteria:

* rheumatoid arthritis,
* legal incompetent patients,
* patients already included in the study for the other hand,
* insufficient knowledge of the German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Michigan Hand Questionnaire - pain subscale | 12 months

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Herren, Dr., Principal Investigator — Department of Handsurgery; Miriam Marks, MSc., Study Chair — Department of Research and Development
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

REFERENCES:
- [Derived] Marks M, Audige L, Herren DB, Schindele S, Nelissen RG, Vliet Vlieland TP. Measurement properties of the German Michigan Hand Outcomes Questionnaire in patients with trapeziometacarpal osteoarthritis. Arthritis Care Res (Hoboken). 2014 Feb;66(2):245-52. doi: 10.1002/acr.22124. PMID 23982906